CLINICAL TRIAL: NCT02839902
Title: Exploratory Study of the Effects of Omega-3-acid Ethyl Esters on the Lipid and Lipoprotein Profile in the Blood
Acronym: LOTUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TAK-085-4002; U1111-1185-0054 (Other: WHO); JapicCTI-163322 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Results first posted 2019-02-11 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2018-08

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — TAK-085; Omacor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAK-085 4g (Experimental): A dose of 2 g of omega-3-acid ethyl esters (TAK-085) capsule is orally administered immediately after meal twice a daily (totally 4g per a day) for 8 weeks, plus a stable HMG-CoA reductase inhibitor regimen (started ≥4 weeks prior to informed consent) at a consistent dose.
  Interventions: Drug: TAK-085
- Control Group (Experimental): Stable HMG-CoA reductase inhibitor regimen at a consistent dose only.
  Interventions: Other: Not treated with omega-3-acid ethyl esters

INTERVENTIONS:
Drug: TAK-085 — Omega-3-acid ethyl esters (TAK-085) capsule
  Arms: TAK-085 4g
Other: Not treated with omega-3-acid ethyl esters — Not treated with omega-3-acid ethyl esters
  Arms: Control Group

SUMMARY:
The purpose of this study is to explore the effects of 8-week treatment with omega-3-acid ethyl esters on the lipid and lipoprotein profile in the blood in hyperlipidemic patients receiving a HMG-CoA reductase inhibitor by use of HPLC in comparison with the control group of patients not treated with omega-3-acid ethyl esters.

DETAILED DESCRIPTION:
This study was designed to explore the effects of omega-3-acid ethyl esters on the lipid and lipoprotein profile in the blood in hyperlipidemic patients receiving a hydroxymethylglutaryl-coenzyme A (HMG-CoA) reductase inhibitor in comparison with the control group of patients not treated with omega-3-acid ethyl esters in an unblinded manner by use of high performance liquid chromatography (HPLC) using highly-sensitive gel filtration columns, which is a technique for analyzing lipoprotein.

Study participants who gave consent and were assessed as eligible in the eligibility assessment will be stratified by the factors of "fasting triacylglycerol (TG; <300 mg/dL or 300 mg/dL≤) and age (<65 years or 65 years≤) at the start of the screening period" and allocated to either the group treated with omega-3-acid ethyl esters or the group not treated with omega-3-acid ethyl esters (1:1 ratio).

ELIGIBILITY:
Inclusion Criteria:

1. Participants diagnosed as hyperlipidemia.
2. Participants constantly receiving a HMG-CoA reductase inhibitor at a stable dose for at least 4 weeks at the start of the observation period.
3. Participants with fasting TG of 150≤ to <400 mg/dL measured at the start of the observation period at Visit 1 (Week -4).
4. Participants who, in the opinion of the principal investigator or the investigator, are capable of understanding the content of the clinical study and complying with the study protocol requirements.
5. Participants who can provide written informed consent prior to the conduction of the clinical study procedures.
6. Participants aged ≥20 years at the time of informed consent at Visit 1 (Week -4).

Exclusion Criteria:

1. Participants who had clinically significant hemorrhagic disorders (e.g., hemophilia, capillary fragility, gastrointestinal ulcer, urinary tract hemorrhage, hemoptysis, and vitreous hemorrhage) within 24 weeks prior to the start of the observation period, or those who concurrently have the above disorders.
2. Participants who had thyroid disorders (hyperthyroidism or hypothyroidism) within 24 weeks prior to the start of the observation period, those who concurrently have the above disorders, or those who are orally receiving a therapeutic drug for thyroid disorder.
3. Participants in whom the type of HMG-CoA reductase inhibitors was changed within 12 weeks prior to the start of observation period.
4. Participants who received an eicosapentaenoic acid (EPA) preparation or an EPA/docosahexaenoic acid (DHA) preparation (including supplements) within 12 weeks prior to the start of observation period.
5. Participants who started antidyslipidemic agents within 4 weeks prior to the start of observation period.
6. Participants with severe hepatic impairment (e.g., Child-Pugh classification C).
7. Participants who were previously diagnosed as lipoprotein lipase deficiency or apoprotein C-II deficiency.
8. Participants who are concurrently having Cushing's syndrome, uremia, systemic lupus erythematosus (SLE), or serum dysproteinemia.
9. Diabetic participants who are currently receiving thiazolidine or insulin.
10. Participants who are concurrently having hypertension of grade IIINote 1). Note 1: Participants with systolic blood pressure of ≥180 mm Hg or diastolic blood pressure of ≥110 mm Hg regardless of treatment with antihypertensive drugs.
11. Participants who are habitual drinkers drinking an average of over 100 mL per day (expressed in terms of quantity of alcohol), or participants with or with a history of drug abuse or addiction.
12. Pregnant, lactating or postmenopausal women.
13. Participants with a history of hypersensitivity or allergy for omega-3-acid ethyl esters.
14. Participants participating in other clinical studies.
15. Participants assessed ineligible in the study by the principal investigator or the investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-12-27 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (7):
- Japan (7):
  - Noda, Chiba
  - Koga, Ibaragi
  - Moriguchi, Osaka
  - Suita, Osaka
  - Fujimi, Saitama
  - Mitaka, Tokyo
  - Saitama

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 7 investigative sites in Japan, from 27 December 2016 to 30 August 2017.
Pre-assignment Details: Participants with a historical diagnosis of hyperlipidemia who were inadequately controlled while receiving a hydroxymethylglutaryl-coenzyme A (HMG-CoA) reductase inhibitor were enrolled in one of two groups, treatment group with omega-3-acid ethyl esters (TAK-085) 2 grams (g) and treatment group without TAK-085 (Control Group).
Groups:
- TAK-085 4 g: A dose of 2 g of omega-3-acid ethyl esters (TAK-085) capsule was orally administered immediately after a meal twice daily (totally 4g per a day) for 8 weeks, plus a stable HMG-CoA reductase inhibitor regimen (started ≥4 weeks prior to informed consent) at a consistent dose.
Period: Overall Study
Arm/Group | TAK-085 4 g | Control Group
Started | 24 | 29
Completed | 24 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS); FAS was defined as participants who were randomized and received at least one dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAK-085 4 g | Control Group | Total
Number analyzed (Participants) | 24 | 29 | 53
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (11.28) | 62.3 (11.67) | 61.5 (11.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 23 | 29 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Japan | 24 | 29 | 53
Height [Mean (Standard Deviation); unit: Centimeters (cm)] | 168.9 (6.05) | 167.7 (7.55) | 168.2 (6.87)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] | 77.93 (9.784) | 77.13 (12.507) | 77.49 (11.257)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2]
  kg/m^2 | 27.27 (2.791) | 27.39 (3.746) | 27.34 (3.317)
Duration of Hyperlipemia [Mean (Standard Deviation); unit: Years] — Mean duration between start of study and first time of diagnosis of hyperlipemia was reported.
  Years | 11.05 (7.590) | 7.76 (5.847) | 9.25 (6.828)
Frequency of Fish Intake [Count of Participants; unit: Participants] — Participants were asked a question about frequency of consumption of fish and answered from 4 types of the answers; Almost Every Day, About Every 2 Days, About Once or Twice per Week, and Rarely. Reported data were the number of participants who selected from 4 answers.
  Participants
    Almost Every Day | 2 | 4 | 6
    About Every Two Days | 6 | 6 | 12
    About Once or Twice Per Week | 15 | 19 | 34
    Rarely | 1 | 0 | 1
Smoking Classification [Count of Participants; unit: Participants]
  Never smoked | 5 | 9 | 14
  Current smoker | 5 | 7 | 12
  Ex-smoker | 14 | 13 | 27
Drinking habit [Count of Participants; unit: Participants] — Participants who answered Yes or No for a question "Drink Alcohol Almost Every Day?" were reported.
  Participants
    Yes | 7 | 9 | 16
    No | 17 | 20 | 37
Fasting Triglycerides [Mean (Standard Deviation); unit: Milligram (mg)/deciliter (dL)] | 208.0 (74.05) | 214.7 (73.12) | 211.7 (72.91)
Cholesterol Concentration in Small Dense Low Density Lipoprotein (sdLDL) Fraction [Mean (Standard Deviation); unit: mg/dL] | 30.285 (5.9109) | 32.981 (9.1346) | 31.760 (7.8879)
Triglycerides Concentration in sdLDL Fraction [Mean (Standard Deviation); unit: mg/dL] | 6.778 (1.8022) | 7.320 (2.0727) | 7.074 (1.9556)
Free Cholesterol Concentration in sdLDL Fraction [Mean (Standard Deviation); unit: mg/dL] | 8.670 (1.6883) | 9.353 (2.3705) | 9.044 (2.0986)
Phospholipid Concentration in sdLDL Fraction [Mean (Standard Deviation); unit: mg/dL] | 31.526 (5.1749) | 33.860 (7.9633) | 32.803 (6.8824)
Particle Size of LDL(Cholesterol Monitor) [Mean (Standard Deviation); unit: Nanometer (nm)] | 25.712 (0.4301) | 25.681 (0.4087) | 25.695 (0.4148)
Particle Size of LDL (Triglycerides Monitor) [Mean (Standard Deviation); unit: nm] — Population: Population Analysis Description: The number analyzed is the number of participants with data available for analysis.
  nm
    number analyzed (Participants) | 9 | 11 | 20
    (all) | 29.378 (1.0152) | 29.005 (0.8946) | 29.173 (0.9442)
Particle Size of LDL (Free Cholesterol Monitor) [Mean (Standard Deviation); unit: nm] | 25.560 (0.4403) | 25.492 (0.4263) | 25.523 (0.4299)
Particle Size of LDL (Phospholipid Monitor) [Mean (Standard Deviation); unit: nm] | 25.335 (0.4431) | 25.263 (0.3945) | 25.296 (0.4147)

OUTCOME MEASURES:

1. Primary Outcome: Percent Changes From Baseline in Concentration of Major 4 Lipid Constituents in Small Dense Low Density Lipoprotein (sdLDL) Fraction
Description: Major 4 lipid constituents refer to cholesterol, triglycerides, free cholesterol, and phospholipid. The reported data are percent of change from baseline in concentration of the each lipid constituents in sdLDL fraction at Week 4 and Week 8.
Time Frame: Baseline, Week 4 and Week 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | TAK-085 4 g | Control Group
Number analyzed (Participants) | 24 | 29
Percent of Change
  Cholesterol at Week 4 | -6.50 (15.745) | 5.05 (11.401)
  Cholesterol at Week 8 | -12.35 (13.519) | 4.64 (17.845)
  Triglycerides at Week 4 | -2.87 (22.917) | 9.71 (23.437)
  Triglycerides at Week 8 | -6.50 (22.615) | 2.74 (20.317)
  Free Cholesterol at Week 4 | -6.32 (12.483) | 2.14 (14.048)
  Free Cholesterol at Week 8 | -6.94 (16.639) | 3.42 (14.516)
  Phospholipid at Week 4 | -8.31 (11.396) | 2.10 (11.297)
  Phospholipid at Week 8 | -10.37 (13.919) | 1.09 (13.440)
Statistical Analysis 1: Comparison: TAK-085 4 g vs Control Group; The least square (LS) mean percentage change was compared between treatment groups with cholesterol concentration in sd LDL fraction at Week 8 using an ANCOVA model; Test type: Other — Least square (LS) mean difference; p = 0.0004, ANCOVA; Least square (LS) mean difference = -17.147, 95% CI 2-sided [-26.344 to -7.950] — TAK-085 4 g - Control Group
Statistical Analysis 2: Comparison: TAK-085 4 g vs Control Group; The least square (LS) mean percentage change was compared between treatment groups with triglycerides concentration in sd LDL fraction at Week 8 using an ANCOVA model; Test type: Other — Least square (LS) mean difference; p = 0.1141, ANCOVA; Least square (LS) mean difference = -9.774, 95% CI 2-sided [-21.986 to 2.439] — TAK-085 4 g - Control Group
Statistical Analysis 3: Comparison: TAK-085 4 g vs Control Group; The least square (LS) mean percentage change was compared between treatment groups with free cholesterol concentration in sd LDL fraction at Week 8 using an ANCOVA model; Test type: Other — Least square (LS) mean difference; p = 0.0248, ANCOVA; Least square (LS) mean difference = -10.246, 95% CI 2-sided [-19.143 to -1.349] — TAK-085 4 g - Control Group
Statistical Analysis 4: Comparison: TAK-085 4 g vs Control Group; The least square (LS) mean percentage change was compared between treatment groups with phospholipid concentration in sd LDL fraction at Week 8 using an ANCOVA model; Test type: Other — Least square (LS) mean difference; p = 0.0047, ANCOVA; Least square (LS) mean difference = -11.511, 95% CI 2-sided [-19.340 to -3.682] — TAK-085 4 g - Control Group

2. Primary Outcome: Percent Changes From Baseline in Triglycerides (TG) to Cholesterol Ratio in sdLDL Fraction
Description: Reported data are percent of change from baseline in in TG to cholesterol ratio in sdLDL fraction at Week 4 and Week 8.
Time Frame: Baseline, Week 4, and Week 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | TAK-085 4 g | Control Group
Number analyzed (Participants) | 24 | 29
Percent of Change
  Week 4 | 4.48 (21.423) | 5.66 (25.908)
  Week 8 | 8.64 (31.398) | -0.94 (17.267)
Statistical Analysis 1: Comparison: TAK-085 4 g vs Control Group; The least square (LS) mean percentage change was compared between treatment groups with TG to cholesterol ratio in sd LDL fraction at Week 8 using an ANCOVA model; Test type: Other — Least square (LS) mean difference; p = 0.1826, ANCOVA; Least square (LS) mean difference = 9.499, 95% CI 2-sided [-4.623 to 23.622] — TAK-085 4 g - Control Group

3. Primary Outcome: Percent Change From Baseline in Mean Particle Sizes of Small Dense Low Density Lipoprotein-cholesterol (sdLDL-C) and Low Density Lipoprotein-cholesterol (LDL-C) Monitored by Major 4 Lipid Constituents
Description: Reported data are percent of change from baseline in mean particle sizes of sdLDL-C and LDL-C monitored by major 4 lipid constituents (cholesterol, triglycerides, free cholesterol, and phospholipid) at Week 4 and Week 8. Here the data were consolidated from results of the two outcome measures ("Change in mean particle sizes of sdLDL-C" and "Change in mean particle sizes of LDL-C") on initial registration information (see History of Change of registration) because sdLDL-C refers to LDL-C which is smaller particle size and heavier density.
Time Frame: Baseline, Week 4, and Week 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | TAK-085 4 g | Control Group
Number analyzed (Participants) | 24 | 29
Percent of Change
  Week 4 (Cholesterol Monitor) | 0.56 (1.217) | -0.39 (0.820)
  Week 8 (Cholesterol Monitor) | 0.99 (1.192) | -0.08 (1.274)
  Week 4 (Triglycerides Monitor): number analyzed (Participants) | 8 | 6
  Week 4 (Triglycerides Monitor) | 0.87 (6.026) | -0.06 (1.367)
  Week 8 (Triglycerides Monitor): number analyzed (Participants) | 5 | 6
  Week 8 (Triglycerides Monitor) | 2.11 (2.715) | 0.52 (3.155)
  Week 4 (Free Cholesterol Monitor) | 0.79 (1.247) | -0.16 (0.953)
  Week 8 (Free Cholesterol Monitor) | 0.90 (1.407) | 0.07 (1.361)
  Week 4 (Phospholipid Monitor) | 0.63 (1.464) | -0.23 (1.018)
  Week 8 (Phospholipid Monitor) | 0.99 (1.316) | 0.09 (1.431)
Statistical Analysis 1: Comparison: TAK-085 4 g vs Control Group; The least square (LS) mean percentage change was compared between treatment groups with particle size (nm) of LDL at Week 8 monitored by cholesterol using an ANCOVA model; Test type: Other — Least square (LS) mean difference; p = 0.0040, ANCOVA; Least square (LS) mean difference = 1.066, 95% CI 2-sided [0.356 to 1.776] — TAK-085 4 g - Control Group
Statistical Analysis 2: Comparison: TAK-085 4 g vs Control Group; The least square (LS) mean percentage change was compared between treatment groups with particle size (nm) of LDL at Week 8 monitored by triglycerides using an ANCOVA model; Test type: Other — Least square (LS) mean difference; p = 0.4428, ANCOVA; Least square (LS) mean difference = 1.553, 95% CI 2-sided [-2.884 to 5.991] — TAK-085 4 g - Control Group
Statistical Analysis 3: Comparison: TAK-085 4 g vs Control Group; The least square (LS) mean percentage change was compared between treatment groups with particle size (nm) of LDL at Week 8 monitored by free cholesterol using an ANCOVA model; Test type: Other — Least square (LS) mean difference; p = 0.0570, ANCOVA; Least square (LS) mean difference = 0.760, 95% CI 2-sided [-0.024 to 1.544] — TAK-085 4 g - Control Group
Statistical Analysis 4: Comparison: TAK-085 4 g vs Control Group; The least square (LS) mean percentage change was compared between treatment groups with particle size (nm) of LDL at Week 8 monitored by phospholipid using an ANCOVA model; Test type: Other — Least square (LS) mean difference; p = 0.0360, ANCOVA; Least square (LS) mean difference = 0.838, 95% CI 2-sided [0.057 to 1.620] — TAK-085 4 g - Control Group

4. Secondary Outcome: Percent Changes From Baseline in Concentration of Major 4 Lipid Constituents in Chylomicron (CM) Fraction
Description: Major 4 lipid constituents refer to cholesterol, triglycerides, free cholesterol, and phospholipid. The reported data are percent of change from baseline in concentration of the each lipid constituents in CM fraction at Week 4 and Week 8.
Time Frame: Baseline, Week 4 and Week 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | TAK-085 4 g | Control Group
Number analyzed (Participants) | 24 | 29
Percent of Change
  Cholesterol at Week 4 | -38.03 (53.008) | 47.42 (149.946)
  Cholesterol at Week 8 | -32.92 (60.170) | -0.68 (65.088)
  Triglycerides at Week 4 | -37.22 (49.604) | 42.62 (132.804)
  Triglycerides at Week 8 | -33.32 (52.994) | -3.74 (55.812)
  Free Cholesterol at Week 4 | -38.13 (50.570) | 60.20 (189.062)
  Free Cholesterol at Week 8 | -30.33 (65.974) | 2.37 (71.895)
  Phospholipid at Week 4 | -40.25 (61.678) | 48.94 (118.843)
  Phospholipid at Week 8 | -38.00 (64.130) | 1.15 (92.004)

5. Secondary Outcome: Percent Changes From Baseline in Concentration of Major 4 Lipid Constituents in Very Low-density Lipoprotein (VLDL) Fraction
Description: Major 4 lipid constituents refer to cholesterol, triglycerides, free cholesterol, and phospholipid. The reported data are percent of change from baseline in concentration of the each lipid constituents in VLDL Fraction at Week 4 and Week 8.
Time Frame: Baseline, Week 4 and Week 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | TAK-085 4 g | Control Group
Number analyzed (Participants) | 24 | 29
Percent of Change
  Cholesterol at Week 4 | -10.45 (17.089) | 5.45 (15.255)
  Cholesterol at Week 8 | -15.16 (19.449) | 1.03 (14.717)
  Triglycerides at Week 4 | -15.21 (23.536) | 7.24 (28.285)
  Triglycerides at Week 8 | -17.26 (24.705) | -1.32 (20.084)
  Free Cholesterol at Week 4 | -13.06 (19.539) | 6.99 (20.379)
  Free Cholesterol at Week 8 | -16.48 (24.694) | 0.64 (17.034)
  Phospholipid at Week 4 | -13.78 (19.839) | 5.99 (19.193)
  Phospholipid at Week 8 | -16.49 (22.717) | -1.09 (16.446)

6. Secondary Outcome: Percent Changes From Baseline in Concentration of Major 4 Lipid Constituents in Low-density Lipoprotein (LDL) Fraction
Description: Major 4 lipid constituents refer to cholesterol, triglycerides, free cholesterol, and phospholipid. The reported data are percent of change from baseline in concentration of the each lipid constituents in LDL Fraction at Week 4 and Week 8.
Time Frame: Baseline, Week 4 and Week 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | TAK-085 4 g | Control Group
Number analyzed (Participants) | 24 | 29
Percent of Change
  Cholesterol at Week 4 | -4.40 (10.300) | 1.44 (11.146)
  Cholesterol at Week 8 | -6.25 (12.087) | 3.45 (11.789)
  Triglycerides at Week 4 | 0.38 (13.307) | 3.82 (10.813)
  Triglycerides at Week 8 | -2.28 (15.034) | 2.19 (12.348)
  Free Cholesterol at Week 4 | -0.37 (12.581) | 0.30 (13.908)
  Free Cholesterol at Week 8 | -0.48 (15.395) | 3.32 (12.404)
  Phospholipid at Week 4 | -3.94 (8.257) | 0.29 (9.809)
  Phospholipid at Week 8 | -4.80 (10.561) | 1.58 (9.817)

7. Secondary Outcome: Percent Changes From Baseline in Concentration of Major 4 Lipid Constituents in High-density Lipoprotein (HDL) Fraction
Description: Major 4 lipid constituents refer to cholesterol, triglycerides, free cholesterol, and phospholipid. The reported data are percent of change from baseline in concentration of the each lipid constituents in HDL Fraction at Week 4 and Week 8.
Time Frame: Baseline, Week 4 and Week 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | TAK-085 4 g | Control Group
Number analyzed (Participants) | 24 | 29
Percent of Change
  Cholesterol at Week 4 | -1.49 (7.316) | 0.64 (8.039)
  Cholesterol at Week 8 | -3.24 (9.567) | 1.48 (8.249)
  Triglycerides at Week 4 | -9.07 (23.323) | 6.20 (23.726)
  Triglycerides at Week 8 | -6.99 (34.397) | 0.91 (19.979)
  Free Cholesterol at Week 4 | -2.56 (9.832) | 3.29 (9.708)
  Free Cholesterol at Week 8 | -3.31 (12.969) | 5.61 (12.174)
  Phospholipid at Week 4 | -6.47 (7.169) | -2.32 (8.029)
  Phospholipid at Week 8 | -6.45 (10.432) | -3.40 (10.212)

8. Secondary Outcome: Percent Changes From Baseline in Concentration of Fatty Acids in Total Lipids
Description: Fatty acids refer to the following 24 acids; Lauric acid, Myristic acid, Myristoleic acid, Palmitic acid, Palmitoleic acid, Stearic acid, Oleic acid, Linoleic acid, Gamma-linolenic acid, Linolenic acid, Arachic acid, Eicosenoic acid, Eicosadienoic acid, 5-8-11 Eicosatrienoic acid, Dihomo-gamma-linolenic acid, Arachidonic acid, Eicosapentaenoic acid, Behenic acid, Erucic acid, Docosatetraenoic acid, Docosapentaenoic acid, Lignoceric acid, Docosahexaenoic acid, and Nervonic acid. The reported data are percent of change from baseline in concentration of these fatty acids in total lipids at Week 4 and Week 8.
Time Frame: Baseline, Week 4 and Week 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | TAK-085 4 g | Control Group
Number analyzed (Participants) | 24 | 29
Percent of Change
  Lauric Acid at Week 4 | -13.26 (56.101) | 50.65 (86.467)
  Lauric Acid at Week 8 | 6.84 (85.494) | 34.60 (138.684)
  Myristic Acid at Week 4 | -21.37 (26.046) | 24.68 (54.142)
  Myristic Acid at Week 8 | -13.31 (33.571) | 5.96 (32.534)
  Myristoleic Acid at Week 4 | -31.40 (25.830) | 32.50 (77.309)
  Myristoleic Acid at Week 8 | -8.54 (100.145) | -0.55 (37.180)
  Palmitic Acid at Week 4 | -12.49 (20.682) | 5.77 (17.277)
  Palmitic Acid at Week 8 | -9.62 (22.355) | -2.63 (15.549)
  Palmitoleic Acid at Week 4 | -22.35 (22.371) | 5.53 (29.987)
  Palmitoleic Acid at Week 8 | -19.25 (27.584) | -1.17 (22.775)
  Stearic Acid at Week 4 | -4.74 (22.322) | 4.03 (16.408)
  Stearic Acid at Week 8 | -3.17 (24.102) | 0.12 (14.957)
  Oleic Acid at Week 4 | -17.77 (23.295) | 3.28 (19.641)
  Oleic Acid at Week 8 | -13.77 (25.958) | -4.90 (15.856)
  Linoleic Acid at Week 4 | -10.47 (17.286) | 2.93 (12.616)
  Linoleic Acid at Week 8 | -11.84 (16.303) | -0.33 (14.748)
  Gamma-linolenic Acid at Week 4 | -34.84 (17.846) | 7.82 (35.906)
  Gamma-linolenic Acid at Week 8 | -35.21 (19.170) | -1.63 (23.426)
  Linolenic Acid at Week 4 | -9.50 (26.598) | 12.09 (34.208)
  Linolenic Acid at Week 8 | -7.27 (30.301) | -0.50 (25.026)
  Arachic Acid at Week 4 | -15.59 (32.158) | 8.20 (35.594)
  Arachic Acid at Week 8 | -7.11 (43.510) | 2.01 (32.969)
  Eicosenoic Acid at Week 4 | -22.66 (30.315) | 6.82 (41.150)
  Eicosenoic Acid at Week 8 | -19.43 (28.872) | 0.80 (27.505)
  Eicosadienoic Acid at Week 4 | -23.82 (18.803) | 0.31 (14.078)
  Eicosadienoic Acid at Week 8 | -21.50 (21.967) | -3.17 (18.978)
  5-8-11 Eicosatrienoic Acid at Week 4 | -42.51 (23.478) | 17.71 (68.061)
  5-8-11 Eicosatrienoic Acid at Week 8 | -48.16 (24.514) | 13.24 (38.481)
  Dihomo-gamma-linolenic Acid at Week 4 | -38.14 (15.452) | 0.89 (17.847)
  Dihomo-gamma-linolenic Acid at Week 8 | -37.18 (15.933) | 1.98 (22.295)
  Arachidonic Acid at Week 4 | -16.23 (11.911) | -1.97 (13.223)
  Arachidonic Acid at Week 8 | -18.35 (14.448) | -2.37 (13.220)
  Eicosapentaenoic Acid at Week 4 | 224.30 (155.842) | 16.58 (53.986)
  Eicosapentaenoic Acid at Week 8 | 238.48 (211.242) | 29.05 (83.267)
  Behenic Acid at Week 4 | -3.33 (47.184) | -0.72 (36.672)
  Behenic Acid at Week 8 | -0.41 (48.418) | 4.09 (39.343)
  Erucic Acid at Week 4 | 27.58 (279.981) | 91.40 (214.836)
  Erucic Acid at Week 8 | -18.05 (71.360) | 139.93 (376.748)
  Docosatetraenoic Acid at Week 4 | -36.43 (17.765) | 4.94 (23.847)
  Docosatetraenoic Acid at Week 8 | -37.74 (17.764) | 1.07 (21.927)
  Docosapentaenoic Acid at Week 4 | 18.16 (27.789) | 5.83 (22.423)
  Docosapentaenoic Acid at Week 8 | 19.89 (33.735) | 5.78 (25.442)
  Lignoceric Acid at Week 4 | -9.06 (20.062) | -2.00 (20.004)
  Lignoceric Acid at Week 8 | -5.01 (25.548) | -2.33 (24.698)
  Docosahexaenoic Acid at Week 4 | 30.71 (25.367) | 3.10 (20.643)
  Docosahexaenoic Acid at Week 8 | 34.00 (41.055) | 7.32 (27.833)
  Nervonic Acid Week 4 | -8.61 (14.334) | 5.98 (25.020)
  Nervonic Acid Week 8 | -7.82 (15.480) | 13.04 (29.043)

9. Secondary Outcome: Percent Changes From Baseline in Eicosatrienoic Acid to Arachidonic Acid (T/T) Ratio in Total Lipids
Description: The reported data are percent of change from baseline in T/T ratio in total lipids at Week 4 and Week 8.
Time Frame: Baseline, Week 4 and Week 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | TAK-085 4 g | Control Group
Number analyzed (Participants) | 24 | 29
Percent of Change
  Week 4 | -11.81 (23.814) | 8.62 (35.529)
  Week 8 | -12.50 (22.656) | 12.07 (43.620)

10. Secondary Outcome: Percent Changes From Baseline in Eicosapentaenoic Acid to Arachidonic Acid (EPA/AA) Ratio in Total Lipids
Description: The reported data are percent of change from baseline in EPA/AA ratio in total lipids at Week 4 and Week 8.
Time Frame: Baseline, Week 4 and Week 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | TAK-085 4 g | Control Group
Number analyzed (Participants) | 24 | 29
Percent of Change
  Week 4 | 293.83 (185.305) | 18.98 (47.676)
  Week 8 | 317.31 (212.306) | 31.77 (75.839)

11. Secondary Outcome: Percent Changes From Baseline in Eicosapentaenoic Acid Plus Docosahexaenoic Acid to Arachidonic Acid (EPA+DHA/AA) Ratio in Total Lipids
Description: The reported data are percent of change from baseline in EPA+DHA/AA ratio in total lipids at Week 4 and Week 8.
Time Frame: Baseline, Week 4 and Week 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | TAK-085 4 g | Control Group
Number analyzed (Participants) | 24 | 29
Percent of Change
  Week 4 | 118.68 (57.033) | 8.87 (28.154)
  Week 8 | 132.20 (76.024) | 14.29 (34.060)

12. Secondary Outcome: Percent Changes From Baseline in Docosahexaenoic Acid to Arachidonic Acid (DHA/AA) Ratio in Total Lipids
Description: The reported data are percent of change from baseline in DHA/AA ratio in total lipids at Week 4 and Week 8.
Time Frame: Baseline, Week 4 and Week 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | TAK-085 4 g | Control Group
Number analyzed (Participants) | 24 | 29
Percent of Change
  Week 4 | 57.80 (31.135) | 6.22 (22.634)
  Week 8 | 66.11 (43.927) | 10.29 (25.525)

13. Secondary Outcome: Change From Baseline in Mean Concentration of sd LDL-C in Total Lipids
Description: There were no reporting data for this outcome measure because the data of change in mean concentration of sdLDL-C in total lipids were not collected and analyzed in this study finally. So here the data input for this outcome measure are NA for each arm.
Time Frame: Baseline, Week 4 and Week 8
Population: There were no reporting data for this outcome measure because the data of change in mean concentration of sdLDL-C in total lipids were not collected and analyzed in this study finally.
Arm/Group | TAK-085 4 g | Control Group
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Percent Change From Baseline in Concentration of Lipids in the Blood
Description: Lipids on this outcome measure include Total cholesterol, Triacylglycerol (TG), HDL-C, non-HDL, and Remnant lipoprotein cholesterol (RemL-C). Reported data are percent of change in concentration of these lipids in the blood at Week 4 and Week 8.
Time Frame: Baseline, Week 4 and Week 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | TAK-085 4 g | Control Group
Number analyzed (Participants) | 24 | 29
Percent of Change
  Total Cholesterol at Week 4 | -5.74 (7.680) | 2.07 (8.336)
  Total Cholesterol at Week 8 | -7.07 (8.325) | 1.43 (8.267)
  TG at Week 4 | -16.57 (27.101) | 9.60 (34.407)
  TG at Week 8 | -14.51 (32.860) | -2.49 (22.313)
  HDL-C (Direct) at Week 4 | -0.36 (8.290) | 0.70 (9.386)
  HDL-C (Direct) at Week 8 | -1.42 (10.575) | 1.16 (8.305)
  Non-HDL at Week 4 | -7.71 (10.152) | 2.65 (9.978)
  Non-HDL at Week 8 | -9.30 (11.473) | 2.07 (10.898)
  RemL-C at Week 4 | -26.62 (29.222) | 15.84 (47.272)
  RemL-C at Week 8 | -26.07 (38.146) | -4.89 (27.442)

15. Secondary Outcome: Percent Change From Baseline in Concentration of Apolipoproteins in the Blood
Description: Apolipoproteins on this outcome measure include Apolipoprotein AI, AII, B, B-48, B-100, CII, CIII, CII/III, and E. Reported data are percent of change in concentration of these apolipoproteins in the blood at Week 4 and Week 8.
Time Frame: Baseline, Week 4 and Week 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | TAK-085 4 g | Control Group
Number analyzed (Participants) | 24 | 29
Percent of Change
  Apolipoprotein AI at Week 4 | -2.54 (5.068) | 1.39 (5.226)
  Apolipoprotein AI at Week 8 | -4.25 (7.541) | 0.30 (6.540)
  Apolipoprotein AII at Week 4 | -6.56 (6.117) | 2.72 (7.886)
  Apolipoprotein AII at Week 8 | -8.17 (7.326) | 2.86 (8.773)
  Apolipoprotein B at Week 4 | -3.48 (7.515) | 2.14 (8.674)
  Apolipoprotein B at Week 8 | -6.57 (9.763) | 1.63 (8.054)
  Apolipoprotein B-48 at Week 4 | -10.38 (41.138) | 39.56 (84.921)
  Apolipoprotein B-48 at Week 8 | -20.50 (35.739) | 28.49 (71.554)
  Apolipoprotein B-100 at Week 4 | -8.30 (13.124) | 0.79 (9.067)
  Apolipoprotein B-100 at Week 8 | -9.09 (13.453) | 2.39 (14.516)
  Apolipoprotein CII at Week 4 | -11.69 (15.395) | 8.07 (16.006)
  Apolipoprotein CII at Week 8 | -17.80 (17.579) | 6.04 (21.676)
  Apolipoprotein CIII at Week 4 | -7.29 (15.338) | 7.57 (15.115)
  Apolipoprotein CIII at Week 8 | -12.14 (15.585) | 3.01 (16.661)
  Apolipoprotein CII/III at Week 4 | -4.02 (13.076) | 1.58 (18.066)
  Apolipoprotein CII/III at Week 8 | -6.02 (14.231) | 3.36 (16.356)
  Apolipoprotein E at Week 4 | -1.57 (19.222) | 4.38 (15.518)
  Apolipoprotein E at Week 8 | -4.24 (18.788) | 0.30 (13.578)

16. Secondary Outcome: Percent Change From Baseline in Lipoprotein Particle Numbers in the Blood
Description: Reported data were percent of changes from baseline in lipoprotein particle numbers in the blood for 4 fractions (CM, VLDL, LDL, and HDL fractions). Data for this outcome measure was reported instead of the outcome measure title of "Change from Baseline in particle number of lipids, apoprotein and lipoprotein" on registration module (see History of Change of registration).
Time Frame: Baseline, Week 4 and Week 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | TAK-085 4 g | Control Group
Number analyzed (Participants) | 24 | 29
Percent of Change
  CM Fraction at Week 4 | -37.40 (50.191) | 42.88 (134.849)
  CM Fraction at Week 8 | -33.40 (54.049) | -3.70 (56.198)
  VLDL Fraction at Week 4 | -6.20 (16.087) | 5.29 (14.765)
  VLDL Fraction at Week 8 | -9.88 (17.551) | 2.37 (13.808)
  LDL Fraction at Week 4 | -4.58 (10.413) | 2.39 (9.059)
  LDL Fraction at Week 8 | -7.43 (9.993) | 3.07 (11.430)
  HDL Fraction at Week 4 | -4.31 (5.517) | 1.80 (5.893)
  HDL Fraction at Week 8 | -6.33 (6.567) | 1.37 (7.687)

ADVERSE EVENTS:
Time Frame: Up to Week 8
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-085 4 g | Control Group
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/29
Other Adverse Events (participants affected / at risk) | 2/24 | 0/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-085 4 g (N=24) | Control Group (N=29)
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/02/NCT02839902/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/02/NCT02839902/SAP_001.pdf